CLINICAL TRIAL: NCT06341907
Title: Application of MRD Combined With Personalized Vaccine in the Adjuvant Treatment of Postoperative Recurrence Prevention of Epithelial Ovarian Cancer
Brief Title: Application of MRD Combined With Personalized Vaccine in the Treatment of Postoperative Recurrence Prevention of EOC
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2024-07-107
Record Dates: First submitted 2024-03-14; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoantigen polypeptide vaccine (Experimental): Each patient synthesized 5 to 20 neoantigen peptides and was injected with 1 to 4 injections of 1ml polypeptide-poly-ICLC mixture each time. The first round of immunization was administered subcutaneously on days 1, 4, 8, 15, and 22, and the second round of immunization was administered on days 54 and 84
  Interventions: Biological: Neoantigen polypeptide vaccine

INTERVENTIONS:
Biological: Neoantigen polypeptide vaccine — Completion of polypeptide neoantigen polypeptide vaccine (day 1, 4, 8, 15, 22, 54, and 84)

SUMMARY:
The goal of this clinical trial is as follows:(1) Establish a clinical technical system for ctDNA dynamic monitoring of MRD in postoperative EOC patients, providing a new technical means for postoperative recurrence prevention and monitoring of EOC patients.(2) Establish a clinical technical system for adjuvant treatment of postoperative recurrence prevention for EOC patients with conventional protocols combined with personalized vaccines, so as to provide a new treatment method for postoperative recurrence prevention for EOC patients, with a view to obtaining a better survival prognosis.(3) To establish and improve the prediction process of Neoantigen for ovarian cancer and the in vitro evaluation system of the effectiveness of neoantigen vaccine, achieve independent innovation of tumor neoantigen vaccine treatment technology, and cultivate a group of technical forces to master the development of modern tumor vaccine drugs.(4) The new technology system has been promoted and applied in 5 hospitals in the province.

DETAILED DESCRIPTION:
Establish a clinical technology system for the application of conventional protocol combined with personalized immune regulation diagnosis and treatment technology in the adjuvant treatment of MRD-positive patients after EOC surgery: Enroll MRD-positive patients, conduct tumor tissue specimen sequencing, analyze neoantigens, prepare personalized immune regulation diagnosis and treatment technology, and conduct adjuvant treatment for recurrence prevention and treatment with conventional protocol combined with personalized immune regulation diagnosis and treatment technology. Blood routine, biochemical, immunological, tumor indicators (CA125, HE4, CEA, CA199, etc.), imaging examinations (CT, PET-CT, MRI and ultrasound examinations of the resection site of the primary lesion or metastasis) and survival time (PFS, OS) of the patients were followed up after treatment to evaluate their effectiveness and safety. To analyze the advantages of routine regimen combined with personalized immunomodulatory diagnosis and treatment technology for adjuvant therapy for recurrence prevention in MRD positive patients after EOC.

The new technology system has been promoted and applied in 5 hospitals in the province: it is evaluated and validated by carrying out prospective multi-center clinical studies to guide the continuous optimization of clinical treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage II, III, and IV epithelial ovarian cancer who can be surgically resected and can provide sufficient tumor tissue samples, including paraffin-embedded (FFPE) blocks or fresh sections of formalin-fixed tissue within six months (approved by the organizer only);
2. 18-70 years old;
3. In the judgment of the researcher, be able to comply with the research protocol;
4. Voluntarily join the study and sign the informed consent;
5. Patients should meet the following hematological indicators: neutrophil count ≥1.5×109 /L; Hemoglobin ≥10.0 g/dL; Platelet count ≥100×109 /L; Total bilirubin ≤2× upper limit of normal (ULN); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2× upper limit of normal value (ULN); Creatinine clearance ≥60 ml/min;
6. Expected survival ≥ 3 months;
7. The performance status of the Eastern Cancer Cooperation Group (ECOG) was 0 or 1.
8. Postoperative ctDNA MRD test was positive, routine blood index was negative, imaging was negative.

Exclusion Criteria:

1. The patient has HIV infection, HBV infection, HCV infection, uncontrolled coronary artery disease or asthma, uncontrolled cerebrovascular disease, or other disease that the investigator considers ineligible;
2. Patients with a history of bone marrow or organ transplantation;
3. People with coagulation disorders;
4. Gastrointestinal bleeding or gastrointestinal bleeding tendency;
5. Subjects with immune deficiency diseases or autoimmune diseases;
6. Patients who have received other immunotherapy within 1 month (such as immunotherapy with checkpoint inhibitors, therapeutic antibodies, immune cell therapy, and immune system modulator therapy);
7. People who may be allergic to immunotherapy;
8. The patient is affected by drug abuse, clinical or psychological or social factors that make informed consent or research implementation affected;
9. Pregnant and lactating women;
10. Patients who are participating in or have participated in other clinical trials within 1 month;
11. Any uncertainty affecting the patient's safety or compliance.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | every 3 months after operation up to 24 months
  Objective Response Rate
PFS | every 3 months after operation up to 24 months
  Progression Free Survival
OS | every 3 months after operation up to 24 months
  Overall Survival
CA 125 | every 3 months after operation up to 24 months
  Carbohydrate antigen 125

SECONDARY OUTCOMES:
Safety Index | every 3 months after operation up to 24 months
  Adverse Events; Serious Adverse Events;Drug-related Death;

CONTACTS AND LOCATIONS:
Overall Officials: Ping Duan, Master, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT06341907/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT06341907/ICF_001.pdf